CLINICAL TRIAL: NCT06445023
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Barzolvolimab in Patients With Chronic Spontaneous Urticaria Who Remain Symptomatic Despite H1 Antihistamine Treatment (EMBARQ-CSU1)
Brief Title: A Phase 3 Study of Barzolvolimab in Participants With Chronic Spontaneous Urticaria
Acronym: EMBARQ-CSU1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDX0159-12; 2024-513208-32-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: CDX-0159; barzolvolimab; chronic spontaneous urticaria; CSU; urticaria activity score; itch severity score; hives severity score
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- barzolvolimab 150 mg (Experimental): barzolvolimab given once as a 300 mg subcutaneous injection followed by 150 mg administered every 4 weeks for 52 weeks
  Interventions: Biological: barzolvolimab
- barzolvolimab 300 mg (Experimental): barzolvolimab given once as a 450 mg subcutaneous injection followed by 300 mg administered every 8 weeks for 52 weeks
  Interventions: Biological: barzolvolimab
- Placebo then barzolvolimab 150 mg (Experimental): Placebo injection subcutaneous every 4 weeks for 24 weeks and then barzolvolimab 300 mg followed by 150 mg administered every 4 weeks for 28 weeks.
  Interventions: Biological: barzolvolimab; Biological: Matching placebo
- Placebo then barzolvolimab 300 mg (Experimental): Placebo injection subcutaneous every 4 weeks for 24 weeks and then barzolvolimab 450 mg followed by 300 mg administered every 8 weeks for 28 weeks.
  Interventions: Biological: barzolvolimab; Biological: Matching placebo

INTERVENTIONS:
Biological: barzolvolimab — Subcutaneous Administration
Biological: Matching placebo — Matching placebo Subcutaneous Administration
  Arms: Placebo then barzolvolimab 150 mg; Placebo then barzolvolimab 300 mg

SUMMARY:
The purpose of this study is to establish the efficacy, safety and tolerability of barzolvolimab in adult participants with Chronic Spontaneous Urticaria (CSU) inadequately controlled by non-sedating second generation H1-antihistamines in comparison to placebo.

DETAILED DESCRIPTION:
This is a global, multicenter, randomized, double-blind, parallel group, placebo-controlled phase 3 study investigating the efficacy, safety and tolerability of barzolvolimab in adult participants with Chronic Spontaneous Urticaria (CSU) who are symptomatic despite treatment with non-sedating second generation H1-antihistamines at 1-4 times the locally approved dose.

There is a screening period of up to 4 weeks, followed by a 24-week placebo-controlled treatment period, a 28-week active treatment period where all participants receive barzolvolimab followed by a 16-week treatment free period.

Approximately 915 adult participants (610 in the active arms and 305 in the placebo arm) will be randomly assigned to the treatment arms.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males and females, >/= 18 years of age.
2. Chronic spontaneous urticaria (CSU) >/= 6 months prior to Screening (Visit 1).
3. CSU despite the use of a stable regimen of second generation non-sedating H1-antihistamine as defined by:

   1. The presence of hives for >/= 6 weeks at any time prior to Visit 1 despite the use of non-sedating H1-antihistamines.
   2. Must be on a stable regimen of second generation non-sedating H1-antihistamine for >/= 4 weeks prior to study treatment.
   3. UAS7 of >/= 16 and ISS7 of >/= 8 during the 7 days prior to study treatment.
4. Normal blood counts and liver function tests.
5. Both males and females of child-bearing potential must agree to use highly effective contraceptives during the study and for 150 days after treatment.
6. Willing and able to complete a daily symptom electronic diary and comply with study visits.
7. Participants with and without prior biologic experience are eligible.

Key Exclusion Criteria:

1. Women who are pregnant or nursing.
2. Chronic urticaria whose predominant manifestation is due to CIndU.
3. Other diseases associated with urticaria.
4. Active pruritic skin condition in addition to CSU.
5. Medical condition that would cause additional risk or interfere with study procedures.
6. Known HIV, hepatitis B or hepatitis C infection.
7. Vaccination of a live vaccine within 30 days prior to Screening (Visit 1) (subjects must agree to avoid live vaccinations during the study). Inactivated vaccines are allowed such as seasonal influenza injection or authorized COVID-19 vaccine.
8. History of anaphylaxis.
9. Prior treatment with barzolvolimab.

There are additional criteria that your study doctor will review with you to confirm you are eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 915 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline to Week 12 of UAS7 (Urticaria Activity Score) | From Day 1 (first dose) to Day 85 (Week 12)
  Evaluate efficacy of barzolvolimab on urticaria activity as measured by urticaria activity score (UAS).
  The UAS7 is a simple scoring system to evaluate urticaria signs and symptoms. It is based on scoring wheals (hive severity score) and itch (itch severity score) separately on a scale of 0 (no signs/symptoms) to 3 (intense signs/symptoms) over 7 days. The final score is calculated by adding together the daily scores, which can range from 0 to 6, for 7 days. This results in a maximum total score of 42, and a minimum possible score of 0.

SECONDARY OUTCOMES:
Mean change from baseline to Week 12 of ISS7 (Itch Severity Score) | From Day 1 (first dose) to Day 85 (Week 12)
  The ISS7 and HSS7 combined together make up the UAS7 scoring system to evaluate urticaria signs and symptoms. The ISS7 is the itch severity score for 7 days, the scores range from 0 to 21.
Mean change from baseline to Week 12 of HSS7 (Hives Severity Score) | From Day 1 (first dose) to Day 85 (Week 12)
  The ISS7 and HSS7 combined together make up the UAS7 scoring system to evaluate urticaria signs and symptoms. The HSS7 score is the wheal/hives severity score for 7 days, the scores range from 0 to 21.
Percentage of participants with UAS7 = 0 at Week 12 | From Day 1 (first dose) to Day 85 (Week 12)
  Proportion of participants who achieve complete absence of hives and itch (UAS7 = 0) at Week 12.
Mean change from baseline in UAS7 in participants refractory to omalizumab treatment at Week 12 | From Day 1 (first dose) to Day 85 (Week 12)
  Evaluate efficacy of barzolvolimab on urticaria activity as measured by urticaria activity score (UAS) in participants who did not respond to or did not tolerate omalizumab.
  The UAS7 is a simple scoring system to evaluate urticaria signs and symptoms. It is based on scoring wheals (hive severity score) and itch (itch severity score) separately on a scale of 0 (no signs/symptoms) to 3 (intense signs/symptoms) over 7 days. The final score is calculated by adding together the daily scores, which can range from 0 to 6, for 7 days. This results in a maximum total score of 42, and a minimum possible score of 0.
Proportion of participants with UAS7 = 0 in participants refractory to omalizumab treatment at Week 12 | From Day 1 (first dose) to Day 85 (Week 12)
  Proportion of participants who achieve complete absence of hives and itch (UAS7 = 0) at Week 12 in participants who did not respond to or did not tolerate omalizumab.
Percentage of participants with UAS7 ≤ 6 at Week 12 | From Day 1 (first dose) to Day 85 (Week 12)
  Proportion of participants who achieve control of their urticaria signs and symptoms (UAS7 </=6) at Week 12.
Mean change from baseline in UAS7 at Week 4 | From Day 1 (first dose) to Day 29 (Week 4)
  Evaluate efficacy of barzolvolimab on urticaria activity as measured by urticaria activity score (UAS).
  The UAS7 is a simple scoring system to evaluate urticaria signs and symptoms. It is based on scoring wheals (hive severity score) and itch (itch severity score) separately on a scale of 0 (no signs/symptoms) to 3 (intense signs/symptoms) over 7 days. The final score is calculated by adding together the daily scores, which can range from 0 to 6, for 7 days. This results in a maximum total score of 42, and a minimum possible score of 0.
Mean change from baseline in UAS7 at Week 24 | From Day 1 (first dose) to Day 169 (Week 24)
  Evaluate efficacy of barzolvolimab on urticaria activity as measured by urticaria activity score (UAS).
  The UAS7 is a simple scoring system to evaluate urticaria signs and symptoms. It is based on scoring wheals (hive severity score) and itch (itch severity score) separately on a scale of 0 (no signs/symptoms) to 3 (intense signs/symptoms) over 7 days. The final score is calculated by adding together the daily scores, which can range from 0 to 6, for 7 days. This results in a maximum total score of 42, and a minimum possible score of 0.
Percentage of participants with UAS7 = 0 at Week 24 | From Day 1 (first dose) to Day 169 (Week 24)
  Proportion of participants who achieve complete absence of hives and itch (UAS7 = 0) at Week 24.
Incidence of Treatment-Emergent Adverse Events | From Day 1 (first dose) to Day 477 (Week 68)
  Occurrence of treatment emergent adverse events and serious adverse events during the study.

CONTACTS AND LOCATIONS:
Locations (245):
- United States (64):
  - Cahaba Dermatology Skin Health Center, Birmingham, Alabama
  - Clear Dermatology & Aesthetics Center Scottsdale, Scottsdale, Arizona
  - First OC Dermatology - Fountain Valley, Fountain Valley, California
  - 310 Clinical Research, Inglewood, California
  - Dermatology Research Associates, Los Angeles, California
  - Focus Clinical Research - Los Angeles, Los Angeles, California
  - Cura Clinical Research, Oxnard, California
  - Allergy and Asthma Consultants, Redwood City, California
  - Acclaim Clinical Research, San Diego, California
  - West Dermatology Research Center, San Diego, California
  - Therapeutics Clinical Research, San Diego, California
  - Orso Health, Inc., Torrance, California
  - Integrated Research of Inland, Inc., Upland, California
  - Western States Clinical Research Inc, Wheat Ridge, Colorado
  - Encore Medical Research Boynton Beach, Boynton Beach, Florida
  - Florida Academic Centers Research, Coral Gables, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - GSI Clinical Research, Margate, Florida
  - International Dermatology Research Inc - Miami, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - GCP Global Clinical Professionals, LLC, St. Petersburg, Florida
  - Alliance Clinical Research of Tampa, Tampa, Florida
  - Paradigm Clinical Research Boise, Boise, Idaho
  - Endeavor Health, Skokie, Illinois
  - DS Research - 1005 E. Lewis & Clark Pkwy Indiana Location, Clarksville, Indiana
  - Dawes Fretzin Clinical Research Group-7910 N Shadeland Ave, Indianapolis, Indiana
  - DS Research of Kentucky, LLC, Louisville, Kentucky
  - Allergy and Asthma Specialists PSC, Owensboro, Kentucky
  - Clinical Trials Management LLC - Southshore Office, Metairie, Louisiana
  - Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland
  - DermAssociates, LLC, Rockville, Maryland
  - Institute For Asthma and Allergy, Wheaton, Maryland
  - David Fivenson MD Dermatolgy PLLC, Ann Arbor, Michigan
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - Resp Medicine Research Institute of MI, Ypsilanti, Michigan
  - Dermatolgy and Skin Cancer Center, Lee's Summit, Missouri
  - MediSearch, LLC, Saint Joseph, Missouri
  - Montana Medical Research, Missoula, Montana
  - Excel Clinical Research - Las Vegas, Las Vegas, Nevada
  - Allergy Partners of N.J., P.C., Ocean City, New Jersey
  - Finger Lakes Medical Research, PLLC, Cortland, New York
  - Sadick Research Group, New York, New York
  - Bexley Dermatology Research, Bexley, Ohio
  - Apex Clinical Research, Canton, Ohio
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Wright State Physicians, Fairborn, Ohio
  - Auni Allergy, Findlay, Ohio
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - Southern Plains Medical Center - Chickasha, Oklahoma City, Oklahoma
  - Allergy Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Portland Allergy and Asthma, Clackamas, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - Clinical Research Philadelphia, LLC, Philadelphia, Pennsylvania
  - National Allergy and Asthma Research, LLC - CRN - PPDS, North Charleston, South Carolina
  - Alina Clinical Trials, Dallas, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Epic Clinical Research, Lewisville, Texas
  - VAST Clinical Research - Plano, Plano, Texas
  - STAAMP Research, LLC - CRN, San Antonio, Texas
  - Allergy and Asthma Care of Waco, Waco, Texas
  - University of Utah - MidValley Dermatology - PPDS, Murray, Utah
  - Premier Clinical Research, Spokane, Washington
- Argentina (16):
  - Buenos Aires Skin, Buenos Aires, Buenos Aires
  - Fundacion Cidea, Buenos Aires, Buenos Aires
  - CEMLO:Centro de Especialidades Medicas Lobos, Lobos, Buenos Aires
  - Hospital Italiano De Buenos Aires, Buenos Aires, Buenos Aires F.D.
  - Conexa Investigacion Clinica, CABA, Buenos Aires F.D.
  - Aprillus Asistencia e Investigacion, CABA, Buenos Aires F.D.
  - CARE- Centro de Alergia y Enfermedades Respiratorias, CABA, Buenos Aires F.D.
  - Centro Respiratorio Infantil, Rosario, Sante Fe
  - Instituto de Especialidades de Salud Rosario, Rosario, Sante Fe
  - Servicio de Investigacion de Patologias Alergicas, Rosario, Sante Fe
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario, Sante Fe
  - C.I.C.E 9 de Julio - Sanatorio 9 de Julio S.A., San Miguel de Tucumán, Tucumán Province
  - Clinica Mayo, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - Centro Médico Vitae, Buenos Aires
  - Instituto de Alergia e Inmunologia del Sur, Buenos Aires
- Belgium (8):
  - UZ Antwerp, Edegem, Antwerpen
  - UZ Leuven, Leuven, Vlaams Brabant
  - UZ Brussel, Brussels
  - Saint Luc, Brussels
  - CHU de Liège, Brussels
  - Hôpital Erasme - Erasme Medical Center - PPDS, Brussels
  - UZ Gent, Ghent
  - Dermatologie Maldegem, Maldegem
- Brazil (11):
  - AlergoAlpha Allergia e Immunologia, Barueri
  - Instituto de Pesquisas Clínicas LTDA Brasilia, Brasília
  - Fundação Universidade de Caxias do Sul - Instituto de Pesquisas em Saúde, Caxias do Sul
  - Centro Paraibano de Pesquisas e Estudos Clínicos, João Pessoa
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul (PUCRS), Porto Alegre
  - Hospital Universitário Clementino Fraga Filho (UFRJ), Rio de Janeiro
  - Clinica IBIS, Salvador
  - Centro de Estudos de Pneumologia da Faculdade de Medecina do ABC, Santo André
  - Centro de Pesquisa SVRI Hospital e Maternidade Christóvão da Gama, Santo André
  - Clínica de Alergia Martti Antila, São Paulo
  - Vidamed Care Clínica E Residência, Vitória
- Bulgaria (11):
  - "Medical center MedTech Services" OOD, Haskovo
  - Diagnostic Consultative Center Pulmed, Plovdiv
  - Aipsimpa D-R Talyat Sali Cholak Eood, Razgrad
  - Medical Center Iskar EOOD, Sofia
  - MC Excelsior OOD, Sofia
  - DCC Fokus - 5 OOD LZIBP, Sofia
  - Medical Center Hera EOOD, Sofia
  - UMHATEM " N.I.Pirogov", Sofia
  - Medical Center Pulmovision, Sofia
  - Medical Center "Zara-Med" EOOD, Stara Zagora
  - MBAL Sv. Panteleymon AD, Yambol
- Canada (8):
  - Alberta DermaSurgery Centre - Probity - PPDS, Edmonton, Alberta
  - Skincare Research, St. John's, Newfoundland and Labrador
  - Triple A Lab, Hamilton, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - Centre for Dermatology and Cosmetic Surgery, Richmond Hill, Ontario
  - Canadian Dermatology Centre - Probity - PPDS, Toronto, Ontario
  - Evidence Based Medical Educator Inc., Toronto, Ontario
  - Rejuvenation Dermatology and Aesthetics, Calgary
- Czechia (4):
  - Fakultní nemocnice Královské Vinohrady, Dermatovenerologická klinika, Prague
  - Sanatorium profesora Arenbergera, Prague
  - Kožní ambulance Fialová, s.r.o., Prague
  - Fakultní nemocnice Bulovka, Dermatovenerologická klinika, Prague
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus N
  - Bispebjerg Hospital, Copenhagen NV
  - Gentofte Hospital, Hellerup
- France (7):
  - Hospices Civils de Lyon - Hôpital Lyon Sud, Pierre-Bénite, Rhone
  - CHU de Grenoble Alpes - Hôpital Michallon, La Tronche
  - Cabinet du Dr Ruer-Mulard Mireille, Martigues
  - CHRU Nantes Hôtel Dieu, Nantes
  - CHU de Nice-Hôpital L'Archet, Nice
  - Hôpital La Pitié Salpêtrière, Paris
  - CHRU Rouen - Hôpital Charles-Nicolle, Rouen
- Germany (11):
  - Praxis Dr. Beate Schwarz, Langenau, Baden-Wurttemberg
  - Rosenpark Research GmbH, Darmstadt, Hesse
  - Siteworks Prüfzentrum Lohne - PPDS, Löhne, Lower Saxony
  - MVZ Dermatologisches Zentrum Bonn GmbH - Praxis Friedensplatz, Bonn, North Rhine-Westphalia
  - ProDerma, Dülmen, North Rhine-Westphalia
  - UKSH Kiel, Kiel, Schleswig-Holstein
  - Medizinisches Versorgungszentrum DermaKiel GmbH, Kiel, Schleswig-Holstein
  - Fraunhofer-Institut für Translationale Medizin und Pharmakologie ITMP - Berlin, Berlin
  - Studienzentrum an der Hase Weyergraf / Frick / Heiber GbR, Bramsche
  - Dermatologie Quist, Mainz
  - LMU Klinikum der Universität München, München
- Greece (4):
  - Naval Hospital of Athens, Athens
  - Andreas Syggros Hospital, Athens
  - Attikon General University Hospital, Attiki
  - General Hospital of Thessaloniki 'Papageorgiou', Thessaloniki
- Italy (6):
  - Azienda Ospedaliero Universitaria delle Marche, Ancona
  - ASST Carlo Poma, Mantova
  - Istituti Clinici Scientifici Maugeri IRCCS, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
  - Centro Ricerche Cliniche Verona s.r.l./Ospedale G.B. Rossi Borgo Roma, Verona
- Malaysia (5):
  - Hospital Pulau Pinang, George Town
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching
- Peru (4):
  - Clinica Internacional - Sede Lima, Lima
  - Clinica Ricardo Palma, Lima
  - Clinica San Felipe, Lima
  - Medic Ser S.A.C. Auna Clinica Delgado, Lima
- Poland (26):
  - NZOZ Specjalistyczny Ośrodek Dermatologiczny "DERMAL", Bialystok
  - Prywatna Praktyka Lekarska Gabinet Pediatryczno-Alergologiczny Anna Ploszczuk, Bialystok
  - Pratia Bydgoszcz, Bydgoszcz
  - Ambulatorium Sp. zo.o., Elblag
  - Centrum Badan Klinicznych PI-House Sp. z o.o, Gdansk
  - "SYNEXUS POLSKA" sp. z o.o. Odział w Katowicach, Katowice
  - Centrum Medyczne Katowice - PRATIA - PPDS, Katowice
  - Polimedica PTG Kielce, Kielce
  - Centrum Nowoczesnych Terapii "Dobry Lekarz" Sp. o.o., Krakow
  - Santa Familia PTG Łódź, Lodz
  - Oddzial Kliniczny Chorob Wewnetrznych, Astmy i Alergii z Odcinkiem dla Dzieci, Uniwesytecki Szpital Kliniczny nr 1 im. N. Barlickiego w Lodzi, Lodz
  - Pratia S.A. Centrum Medyczne Pratia Poznań, Poznan
  - Specjalistyczna Przychodnai Lekarska Alergo-Med Sp. z o.o., Poznan
  - Synexus Polska Sp. z o.o. - Poznaniu, Poznan
  - NSZOZ Puls-Med Anna Bogusz, Agnieszka Musielak spolka jawna, Skarżysko-Kamienna
  - Laser Clinic S.C, Szczecin
  - MICS Centrum Medyczne Torun, Torun
  - Klinika Ambroziak Dermatologia, Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - FutureMeds - Targowek - PPDS, Warsaw
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. Prof. Dr hab. Med. Eleonory Reicher, Warsaw
  - Ginemedica, Wroclaw
  - Diagnostic Consultative Center Pulmed, Wroclaw
  - Przychodnia FutureMeds Wroclaw, Wroclaw
  - EuroMediCare Szpital Specjalistyczny z Przychodnia we Wroclawiu, Wroclaw
  - Slaski Park Technologii Medycznych Kardio-Med Silesia Sp. z o. o., Zabrze
- Portugal (9):
  - ULS da Região de Aveiro, EPE - Hospital Infante D. Pedro, Aveiro
  - Centro Clínico Académico, Braga - Hospital de Braga, Braga
  - ULS de Coimbra, EPE - Hospitais da Universidade de Coimbra, Coimbra
  - Hospital Lusiadas Lisboa, Lisbon
  - Unidade Local de Saúde de Santa Maria, Lisbon
  - ULS de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - ULS de Santo António, EPE - Hospital de Santo António, Porto
  - ULS da Arrábida, EPE - Hospital de São Bernardo, Setúbal
  - Unidade Local de Saúde de Gaia/Espinho - Unidade I, Vila Nova de Gaia
- South Africa (14):
  - Iatros International, Bloemfontein, Free State
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - Ubuntu Clinical Research, Krugersdorp, Gauteng
  - Newtown Clinical Research Centre, Newtown, Gauteng
  - About Allergy, Pretoria, Gauteng
  - Ryexo Clinical Research, Pretoria, Gauteng
  - FCRN Clinical Trial Centre, Vereeniging, Gauteng
  - Synapta Clinical Research, Durban, KwaZulu-Natal
  - University of Cape Town Lung Institute, Mowbray, Western Cape
  - Infinity Dermatology Inc, Durban
  - Meditrial, Pietermaritzburg
  - Global Clinical Trials, Pretoria
  - Sandton Medical Research Centre, Sandton
  - Allergy and Asthma Centre, Westville
- South Korea (7):
  - Hanyang University Seoul Hospital, Seongdong, Seoul Teugbyesolsi
  - Korea University Ansan Hospital, Ansan
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Spain (10):
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - C.H. Regional Reina Sofia, Córdoba
  - Future Meds Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Complejo Asistencial Universitario De Salamanca, Salamanca
  - Hospital Universitario de la Plana, Villarreal de Huerva
- Taiwan (10):
  - National Taiwan University Hospital Hsin-Chu Branch, Hsinchu
  - Chang Gung Medical Foundation Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital -PPDS, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - MacKay Memorial Hospital -Taipei branch, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- Turkey (Türkiye) (7):
  - Ankara Universitesi Tip Fakultesi Hastaneleri - Cebeci Hastanesi, Ankara
  - Gazi Universitesi Saglik Arastirma ve Uygulama Merkezi, Ankara
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Fatih
  - Kocaeli Universitesi Tip Fakultesi Hastanesi, Kocaeli
  - Erciyes University School of Medicine, Melikgazi
  - Ondokuz Mayis University Hospital, Samsun
  - Karadeniz Teknik Universitesi Tip Fakultesi Hastanesi, Trabzon

IPD SHARING:
Plan to Share IPD: Undecided